CLINICAL TRIAL: NCT01768572
Title: A Randomized, Double-Blind, Double-Dummy Study Assessing The Safety and Tolerability of Sarilumab and Tocilizumab In Patients With Rheumatoid Arthritis Who Are Inadequate Responders to or Intolerant of TNF Antagonists
Brief Title: To Evaluate The Safety of SAR153191 (REGN88) and Tocilizumab Added to Other RA Drugs in Patients With RA Who Are Not Responding to or Intolerant of Anti-TNF Therapy (SARIL-RA-ASCERTAIN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFY13370; 2012-003536-23; U1111-1133-7839 (Other: UTN)
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; tocilizumab; Hydroxychloroquine; Methotrexate; Sulfasalazine; Leflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sarilumab 150 mg q2w (Experimental): Sarilumab 150 mg subcutaneous (SC) injection once every 2 weeks (q2w) and placebo intravenous (IV) infusion once every 4 weeks (q4w) was added to one or a combination of the nonbiologic disease modifying antirheumatic drug (DMARD), hydroxychloroquine, methotrexate, sulfasalazine and/or leflunomide for 24 weeks, except for the simultaneous use of leflunomide and methotrexate.
  Interventions: Drug: sarilumab SAR153191 (REGN88); Drug: hydroxychloroquine; Drug: methotrexate; Drug: sulfasalazine; Drug: leflunomide; Drug: intravenous placebo
- Sarilumab 200 mg q2w (Experimental): Sarilumab 200 mg SC injection q2w and placebo IV infusion q4w was added to one or a combination of the nonbiologic DMARD, hydroxychloroquine, methotrexate, sulfasalazine and/or leflunomide for 24 weeks, except for the simultaneous use of leflunomide and methotrexate.
  Interventions: Drug: sarilumab SAR153191 (REGN88); Drug: hydroxychloroquine; Drug: methotrexate; Drug: sulfasalazine; Drug: leflunomide; Drug: intravenous placebo
- Tocilizumab q4w (Active Comparator): Tocilizumab 4 mg/kg or 8 mg/kg IV infusion q4w and placebo SC injection q2w was added to one or a combination of the nonbiologic DMARD, hydroxychloroquine, methotrexate, sulfasalazine and/or leflunomide for 24 weeks, except for the simultaneous use of leflunomide and methotrexate.
  Interventions: Drug: tocilizumab; Drug: hydroxychloroquine; Drug: methotrexate; Drug: sulfasalazine; Drug: leflunomide; Drug: subcutaneous placebo

INTERVENTIONS:
Drug: sarilumab SAR153191 (REGN88) — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: Sarilumab 150 mg q2w; Sarilumab 200 mg q2w
Drug: tocilizumab — Pharmaceutical form: solution Route of administration: intravenous
  Arms: Tocilizumab q4w
Drug: hydroxychloroquine — Dispensed according to local practice.
Drug: methotrexate — Dispensed according to local practice.
Drug: sulfasalazine — Dispensed according to local practice.
Drug: leflunomide — Dispensed according to local practice.
Drug: subcutaneous placebo — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: Tocilizumab q4w
Drug: intravenous placebo — Pharmaceutical form: solution Route of administration: intravenous
  Arms: Sarilumab 150 mg q2w; Sarilumab 200 mg q2w

SUMMARY:
Primary Objective:

To assess, in the same study, the safety of sarilumab and tocilizumab in participants with rheumatoid arthritis (RA) who were inadequate responders to or intolerant of tumor necrosis factor (TNF) antagonists.

DETAILED DESCRIPTION:
Total study duration was up to 34 weeks: Screening up to 28 days, treatment phase of 24 weeks, and post-treatment follow-up of 6 weeks.

After completion of the treatment phase of this study, participants were eligible to enter a long term safety study (LTS11210) for active treatment with SAR153191 (REGN88).

ELIGIBILITY:
Inclusion criteria:

Diagnosis of RA was, according to the American College of Rheumatology (ACR)/European League against Rheumatism (EULAR) 2010 Rheumatoid Arthritis Classification Criteria with ≥ 3 months disease duration

ACR Class I-III functional status, was based on the 1991 revised criteria. Moderate-to-severely active RA. Anti-TNF therapy failures, was defined as participants with an inadequate clinical response was defined by the investigator, after being treated for at least 3 consecutive months, and/or intolerance to at least 1 TNF-antagonist, resulting in or requiring their discontinuation. TNF-antagonists were include, but were not limited to, etanercept, infliximab, adalimumab, golimumab and/or certolizumab pegol

Continuous treatment with one or a combination of non-biologic disease modifying antirheumatic drugs (DMARDs) for at least 12 consecutive weeks prior to screening and on a stable dose(s) for at least 6 consecutive weeks prior to screening:

* Methotrexate - 10 to 25 milligram/week orally or parenteral (or per local labelling requirements if the dose range differs)
* Leflunomide - 10 to 20 mg orally daily
* Sulfasalazine (SSZ) - 1000 to 3000 mg orally daily
* Hydroxychloroquine (HCQ) - 200 to 400 mg orally daily

Exclusion criteria:

Participants <18 years of age. Use of parenteral corticosteroids or intra-articular corticosteroids within 4 weeks prior to screening

Use of oral corticosteroids in a dose higher than prednisone 10 mg or equivalent per day, or a change in dosage within 4 weeks prior to screening

Past history of, or current, autoimmune or inflammatory systemic or localized joint disease(s) other than RA

History of juvenile idiopathic arthritis or arthritis onset prior to age 16. Severe systemic RA, including but not limited to vasculitis, pulmonary fibrosis, and/or Felty's syndrome

Participation in any clinical research study that evaluated an investigational drug or therapy within 5 half-lives or 60 days of the Screening Visit, whichever was longer

Participants with active tuberculosis or latent tuberculosis infection. Prior or current history of interstitial lung disease. Prior treatment with anti-interleukin (IL) -6 or anti-IL-6R therapies, including but not limited to tocilizumab or sarilumab

Treatment with anti-TNF agents, as follows:

* Etanercept: within 28 days prior to randomization
* Infliximab, adalimumab, golimumab, certolizumab pegol: within 42 days prior to randomization

Treatment with RA-directed biologic agents with non- TNF-α antagonist mechanisms without adequate washout as follows:

* Anakinra: within 28 days prior to randomization
* Abatacept: within 42 days prior to randomization
* Rituximab or other cell depleting agent: Within 6 months prior to randomization or until total lymphocyte count and CD 19+ lymphocyte count were normalized, or whichever was longer

Prior treatment with a janus kinase (JAK) inhibitor (eg, tofacitinib). Participants with a history of invasive opportunistic infection. Prior or current history of malignancy, including lymphoproliferative diseases, other than adequately-treated carcinoma in-situ of the cervix, nonmetastatic squamous cell or basal cell carcinoma of the skin, within 5 years prior to the randomization (baseline) visit

Prior or current history of other significant concomitant illness(es) that, according to Investigator's judgement, was adversely affect the participant's participation in the study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (78):
- United States (14):
  - Investigational Site Number 840152, Huntsville, Alabama
  - Investigational Site Number 840151, Colorado Springs, Colorado
  - Investigational Site Number 840153, Aventura, Florida
  - Investigational Site Number 840033, Fort Lauderdale, Florida
  - Investigational Site Number 840048, Miami, Florida
  - Investigational Site Number 840155, Palm Harbor, Florida
  - Investigational Site Number 840013, Wheaton, Maryland
  - Investigational Site Number 840154, Boston, Massachusetts
  - Investigational Site Number 840150, Lansing, Michigan
  - Investigational Site Number 840062, Reading, Pennsylvania
  - Investigational Site Number 840038, Austin, Texas
  - Investigational Site Number 840022, Dallas, Texas
  - Investigational Site Number 840156, Dallas, Texas
  - Investigational Site Number 840074, Mesquite, Texas
- Argentina (6):
  - Investigational Site Number 032006, Caba
  - Investigational Site Number 032010, Ramos Mejía
  - Investigational Site Number 032013, Rosario
  - Investigational Site Number 032015, San Fernando
  - Investigational Site Number 032004, San Miguel de Tucumán
  - Investigational Site Number 032005, San Miguel de Tucumán
- Investigational Site Number 056010, Leuven, Belgium
- Brazil (2):
  - Investigational Site Number 076001, Curitiba
  - Investigational Site Number 076030, São José do Rio Preto
- Czechia (3):
  - Investigational Site Number 203009, Liberec
  - Investigational Site Number 203011, Prague
  - Investigational Site Number 203010, Prague
- Estonia (2):
  - Investigational Site Number 233010, Tallinn
  - Investigational Site Number 233002, Tallinn
- Finland (2):
  - Investigational Site Number 246001, Helsinki
  - Investigational Site Number 246010, Riihimäki
- Hungary (6):
  - Investigational Site Number 348014, Budapest
  - Investigational Site Number 348022, Budapest
  - Investigational Site Number 348021, Esztergom
  - Investigational Site Number 348016, Kistarcsa
  - Investigational Site Number 348009, Szolnok
  - Investigational Site Number 348015, Szombathely
- Israel (2):
  - Investigational Site Number 376010, Haifa
  - Investigational Site Number 376011, Tel Aviv
- Italy (2):
  - Investigational Site Number 380002, Florence
  - Investigational Site Number 380005, Genova
- Mexico (5):
  - Investigational Site Number 484008, Durango
  - Investigational Site Number 484035, León
  - Investigational Site Number 484009, Mérida
  - Investigational Site Number 484001, México, D.F.
  - Investigational Site Number 484036, Zapopan
- Netherlands (2):
  - Investigational Site Number 528010, Amsterdam
  - Investigational Site Number 528001, Leiden
- Norway (2):
  - Investigational Site Number 578010, Kristiansand
  - Investigational Site Number 578006, Tønsberg
- Poland (5):
  - Investigational Site Number 616019, Bydgoszcz
  - Investigational Site Number 616054, Bytom
  - Investigational Site Number 616030, Lublin
  - Investigational Site Number 616031, Warsaw
  - Investigational Site Number 616017, Warsaw
- Romania (6):
  - Investigational Site Number 642006, Brăila
  - Investigational Site Number 642021, Bucharest
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642020, Bucharest
  - Investigational Site Number 642010, Bucharest
  - Investigational Site Number 642022, Târgovişte
- Russia (7):
  - Investigational Site Number 643017, Kemerovo
  - Investigational Site Number 643020, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643031, Moscow
  - Investigational Site Number 643030, Moscow
  - Investigational Site Number 643032, Saint Petersburg
- Spain (3):
  - Investigational Site Number 724020, Barcelona
  - Investigational Site Number 724021, Santander
  - Investigational Site Number 724022, Seville
- Sweden (2):
  - Investigational Site Number 752004, Malmo
  - Investigational Site Number 752002, Uppsala
- United Kingdom (6):
  - Investigational Site Number 826004, Doncaster
  - Investigational Site Number 826006, Edinburgh
  - Investigational Site Number 826001, Leeds
  - Investigational Site Number 826002, London
  - Investigational Site Number 826005, Southampton
  - Investigational Site Number 826025, Wigan

REFERENCES:
- [Derived] Rehberg M, Giegerich C, Praestgaard A, van Hoogstraten H, Iglesias-Rodriguez M, Curtis JR, Gottenberg JE, Schwarting A, Castaneda S, Rubbert-Roth A, Choy EHS; MOBILITY, MONARCH, TARGET, and ASCERTAIN investigators. Identification of a Rule to Predict Response to Sarilumab in Patients with Rheumatoid Arthritis Using Machine Learning and Clinical Trial Data. Rheumatol Ther. 2021 Dec;8(4):1661-1675. doi: 10.1007/s40744-021-00361-5. Epub 2021 Sep 14. PMID 34519964
- [Derived] Kovalenko P, Paccaly A, Boyapati A, Xu C, St John G, Nivens MC, Davis JD, Rippley R, DiCioccio AT. Population Pharmacodynamic Model of Neutrophil Margination and Tolerance to Describe Effect of Sarilumab on Absolute Neutrophil Count in Patients with Rheumatoid Arthritis. CPT Pharmacometrics Syst Pharmacol. 2020 Jul;9(7):405-416. doi: 10.1002/psp4.12534. Epub 2020 Jun 20. PMID 32453485
- [Derived] Emery P, Rondon J, Parrino J, Lin Y, Pena-Rossi C, van Hoogstraten H, Graham NMH, Liu N, Paccaly A, Wu R, Spindler A. Safety and tolerability of subcutaneous sarilumab and intravenous tocilizumab in patients with rheumatoid arthritis. Rheumatology (Oxford). 2019 May 1;58(5):849-858. doi: 10.1093/rheumatology/key361. PMID 30590833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 78 centers in 19 countries. A total of 389 participants were screened between 25 March 2013 and 02 April 2014, 187 of whom were screen failures. Screen failures were mainly due to failure to meet inclusion and exclusion criteria.
Pre-assignment Details: Randomization of participants were stratified by region and screening value of absolute neutrophil count. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in 1:1:2 (sarilumab 150 mg q2w: sarilumab 200 mg q2w: tocilizumab q4w). 202 participants were randomized.
Groups:
- Sarilumab 150 mg q2w: Sarilumab 150 mg subcutaneous (SC) injection once every 2 weeks (q2w) and placebo intravenous (IV) infusion once every 4 weeks (q4w) was added to one or a combination of the nonbiologic disease modifying antirheumatic drug (DMARD) for 24 weeks.
- Sarilumab 200 mg q2w: Sarilumab 200 mg SC injection q2w and placebo IV infusion q4w was added to one or a combination of the nonbiologic DMARD for 24 weeks.
- Tocilizumab q4w: Tocilizumab 4 mg/kg or 8 mg/kg IV infusion q4w and placebo SC injection q2w was added to one or a combination of the nonbiologic DMARD for 24 weeks. Dose for tocilizumab could be up-titrated to 8 mg/kg or down-titrated to 4 mg/kg based on clinical response as per Investigator's discretion.
Period: Overall Study
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w | Tocilizumab q4w
Started | 49 | 51 | 102
Completed | 40 | 39 | 96
Not Completed | 9 | 12 | 6
Not completed — Adverse Event | 7 | 8 | 4
Not completed — Lack of Efficacy | 1 | 3 | 1
Not completed — Other, Not due to an adverse event | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sarilumab 150 mg q2w: Sarilumab 150 mg SC injection q2w and placebo IV infusion q4w was added to one or a combination of the nonbiologic DMARD for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w | Tocilizumab q4w | Total
Number analyzed (Participants) | 49 | 51 | 102 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (12.1) | 51.7 (13.1) | 50.4 (13.0) | 51.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 82 | 162
  Male | 8 | 12 | 20 | 40
Duration of rheumatoid arthritis (RA) since diagnosis [Mean (Standard Deviation); unit: years] | 13.59 (8.24) | 10.45 (7.57) | 10.84 (8.91) | 11.41 (8.48)
RA functional class [Number; unit: participants] — RA Class I participants: completely able to perform usual activities of daily living (self-care, vocational and avocational); Class II participants: able to perform usual self-care and vocational activities, but limited in avocational activities; Class III participants: able to perform usual self-care activities, but limited in vocational and avocational activities; Class IV participants: limited in ability to perform usual self-care, vocational and avocational activities.
  participants
    I | 10 | 4 | 16 | 30
    II | 25 | 33 | 62 | 120
    III | 14 | 14 | 24 | 52
    IV | 0 | 0 | 0 | 0
Health Assessment Questionnaire Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — Participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: HAQ-DI is consisted of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; activities are rated on a 4-point scale where 0=best and 3=worst. Overall score was computed as the sum of domain scores and divided by the number of domains answered, ranging from 0 to 3, where 0 = no disability and 3 = very severe, high-dependency disability.
  units on a scale | 1.63 (0.66) | 1.71 (0.60) | 1.78 (0.63) | 1.72 (0.63)
Disease Activity Score for 28 Joints- C-reactive protein (DAS28-CRP) [Mean (Standard Deviation); unit: score on scale] — The DAS28-CRP is a composite score that contains 4 variables: Tender Joints Count (based on 28 joints), Swollen Joints Count (based on 28 joints), general health assessment and high sensitivity C-reactive protein (hs-CRP) in mg/L or erythrocyte sedimentation rate (ESR) in mm/hr. It ranges from 0-10 with a lower score indicating less disease activity. A DAS28-CRP above 5.1 indicates high disease activity, whereas a below 3.2 indicates low disease activity and below 2.6 as disease remission.
  score on scale | 5.85 (0.92) | 5.88 (0.97) | 5.91 (1.01) | 5.89 (0.97)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and does not necessary have to have a causal relationship with treatment. All adverse events that occurred from the first dose of the study drug administration up to 60 days after the end of treatment visit were considered as TEAEs. Serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or a medically important event. A summary of SAEs, all other non-serious AEs, regardless of causality, are reported in AE section.
Time Frame: Up to 211 days
Population: The safety population consisted of all randomized participants who received at least 1 dose or a partial dose of study drug analyzed according to the treatment actually received.
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w | Tocilizumab q4w
Number analyzed (Participants) | 49 | 51 | 102
participants
  Any TEAE | 33 | 36 | 68
  Any treatment-emergent SAE | 1 | 3 | 7
  Any TEAE leading to death | 0 | 0 | 1
  Any TEAE leading to discontinuation | 6 | 8 | 4

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Day 211) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent that is AEs that developed/worsened that occurred during 'TEAE period' (first dose of study drug to last dose of study drug+60 days, last contact date, or the date of death, whichever came first). Analysis was performed on safety population.
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w | Tocilizumab q4w
Serious Adverse Events (participants affected / at risk) | 1/49 | 3/51 | 7/102
Other Adverse Events (participants affected / at risk) | 33/49 | 36/51 | 66/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150 mg q2w (N=49) | Sarilumab 200 mg q2w (N=51) | Tocilizumab q4w (N=102)
Erysipelas (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150 mg q2w (N=49) | Sarilumab 200 mg q2w (N=51) | Tocilizumab q4w (N=102)
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 3 | 4
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 2
Otitis media (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 7
Urinary tract infection (Infections and infestations) | 4 | 1 | 6
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginitis trichomonal (Infections and infestations) | 1 | 0 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 8 | 3
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 4
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 4
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 1
Dark circles under eyes (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 4
Vascular fragility (Vascular disorders) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 1 | 7
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Hand deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 6
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Injection site erythema (General disorders) | 4 | 4 | 1
Injection site macule (General disorders) | 1 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 1
Injection site papule (General disorders) | 0 | 0 | 1
Injection site pruritus (General disorders) | 2 | 1 | 1
Injection site rash (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 2
Nodule (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 5
Blood cholesterol increased (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0
Glomerular filtration rate increased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 3
Neutrophil count increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 3 | 9
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.